CLINICAL TRIAL: NCT07066696
Title: Mindfulness and Compassion Program for the Improvement of Emotional and Behavioral Problems, Academic Performance and School Climate in Students in the Last Cycle of Primary Education (Cuida2 Project)
Brief Title: Mindfulness and Compassion Program for the Improvement of Emotional and Behavioral Problems, Academic Performance and School Climate in Students in the Last Cycle of Primary Education.
Acronym: Cuida2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Mª Teresa Navarro Gil, Principal Investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI24/587
Record Dates: First submitted 2025-06-18; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Mindfulness; Compassion; Self-Compassion; Academic Performance; School Climate; Mental Health; Primary School Students
Keywords: Mindfulness; Compassion; Self-compassion; Primary School Students; Emotional and Behavioural Problems; School Climate; Academic Performance
MeSH Terms: conditions — Psychological Well-Being; Mental Disorders | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cuida2 (Experimental): The "CUIDA2" program is an adaptation of the manual "The practice of compassion. Kindness with others and with oneself" (2019) by Dr. Javier García Campayo. It comprises a total of 9 sessions of approximately 50 minutes (one class). This program is structured in 3 modules: Module I mindfulness, module II compassion and module III convergence of the previous elements. Each module includes group dynamics, short meditation practices adapted to the trainees and the explanation of the main theoretical contents through exercises and stories.
  Interventions: Behavioral: Mindfulness and Compassion Program
- Relaxation (Active Comparator): The active control group consists of a relaxation programme consisting of 9 sessions. The sessions will be given weekly (once a week) and have an estimated duration of 50 minutes. Different breathing practices and exercises and relaxation techniques such as visualisation, Jacobson's progressive relaxation and Schultz's autogenic relaxation will be worked on.
  Interventions: Behavioral: Mindfulness and Compassion Program; Behavioral: Relaxation

INTERVENTIONS:
Behavioral: Mindfulness and Compassion Program — The "CUIDA2" program is an adaptation of the manual "The practice of compassion. Kindness with others and with oneself" (2019) by Dr. Javier García Campayo. It comprises a total of 9 sessions of approximately 50 minutes (one class).
  This program is structured in 3 modules: Module I mindfulness, module II compassion and module III convergence of the previous elements. Each module includes group dynamics, short meditation practices adapted to the trainees and the explanation of the main theoretical contents through exercises and stories.
  Other Names: Cuida2
Behavioral: Relaxation — The active control group is composed of a relaxation program consisting of 9 sessions. The sessions will be given weekly (once a week) and have an estimated duration of 50 minutes. Different breathing practices and exercises and relaxation techniques such as visualization, Jacobson's progressive relaxation and Schultz's autogenic relaxation will be used.
  Arms: Relaxation

SUMMARY:
This randomized controlled trial aims to evaluate the efficacy of a Mindfulness and Compassion program to improve emotional and behavioral problems, academic performance and school climate of students in the last cycle of Primary Education.

Participants will be randomly assigned to the Cuida2 program or to an active control group practicing relaxation.

The different variables studied will be evaluated before and after the intervention, and at a three months follow-up. These evaluations will be carried out by the students and their families. In addition, a qualitative exploration will be carried out at the end of the programs, also including the teachers' perceptions.

DETAILED DESCRIPTION:
In recent years, special interest has been given to the social and emotional development of students due to the high prevalence of mental health problems, low academic motivation, school dropout, bullying and school aggression during late childhood and early adolescence. During this stage, students experience the transition from childhood to adolescence, which entails important biological, neurodevelopmental, social and psychological changes that can be difficult to cope with. The scientific literature indicates that there is a high prevalence of mental health disorders that affect the quality of life in childhood and that, if not adequately treated, can be maintained and aggravated during the adolescent years. On the other hand, data on school coexistence is relevant given the great impact it has on students' academic learning and personal development. As a result, problems related to understanding, respect and care for oneself and others are becoming increasingly important in the school population.

In view of the above, it is important to implement prevention and early intervention strategies that promote the proper overall development of students in order to prevent the effects of behavioural and emotional alterations that could lead to mental and physical health problems during this period of life and provide them with sufficient tools to deal with the various situations that arise in both the academic and personal spheres.

A growing number of studies suggest that Mindfulness-Based Interventions (hereafter MBI) produce numerous benefits such as improved attention, concentration emotional intelligence, self-control and reduced or prevented symptoms of anxiety and depression.

In addition, different studies find that more self-compassionate people experience higher levels of happiness, life satisfaction, emotional intelligence, acceptance and less fear of failure, depression and stress. On an interpersonal level, they show greater social connectedness, more tolerance for the imperfections of others and a greater willingness to help those in need.

The study population is Aragonese learners aged 10-12 years in the 5th and 6th grades of primary school. The total sample size needed has been calculated assuming a moderate effect of the mindfulness and compassion programme versus the control group on the main variable "emotional and behavioural problems" in the post-treatment. With a 1:1 allocation ratio, a statistical power of 80%, a bilateral alpha of 0.05, and a standard effect size d = 0.40 when comparing the two arms, a total of 198 participants (99 per group) were obtained; assuming a 10% drop-out rate at follow-up, the total required sample size was set at approximately 220 participants (about 110 per group to be randomised through the Epidat programme). On the other hand, the participation of a parent or guardian of each pupil will be requested, for a total of 220 family members. Finally, the tutors of each class, around 8 teachers, will be involved.

Variables assessed included emotional and behavioural problems, compassion and academic performance. Assessments will be conducted before and after the intervention, and at a three months follow-up.

Socio-demographic characteristics will be described by means of mean, standard deviation, frequencies and percentages, according to their distribution. Comparisons will be made to verify that there are no differences at baseline, using the t-test and the chi-square test. An analysis of covariance (ANCOVA) will be performed for both the primary measure "Child and Adolescent Assessment System, SENA" and the secondary measures, "CSC and academic achievement" by intention to treat (ITT), on the outcome variables after the intervention and on the follow-up measure. The baseline scores of the corresponding dependent variable, and those socio-demographic factors that show significant differences between the two groups at the first measurement point, will be included as covariates. The effect size will be calculated using the partial eta squared value. Values ≤ 0.01 correspond to a low effect size, = 0.06 to a medium effect size and ≥ 0.14 to a large effect size. Contrasts will be made between the pre-test and post-test measures for each group separately, using the corresponding t-test. The level of significance adopted will be α < 0.05.

To analyse the qualitative data "semi-structured global impression interview" two researchers will independently conduct thematic content analysis on the textual corpus following the constant comparison method (Glaser and Strauss, 1967), and developing an initial list of codes. Discrepancies between codings will be resolved by discussion, adjusting the initial list of codes until a common conceptual name is used. Similar codes will be grouped into a single underlying theme in order to represent a more parsimonious solution, allowing the emerging conceptual structure to gain in density. This latter categorisation will be specifically reviewed for discrepancies, resolving possible disagreements and resulting in a final update of the list of themes.

ELIGIBILITY:
Inclusion Criteria:

* To be a pupil, parent/guardian of a child or minor under guardianship or academic tutor in the 5th or 6th year of Primary Education.
* Fluent in Spanish.
* Provided informed consent.

Exclusion Criteria:

* Participant's decision to withdraw from the study at any point

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 448 (Estimated)
Dates: Start 2025-10-06 (Estimated); Primary Completion 2026-06-20 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Child and Adolescent Assessment System (Acronym in Spanish: SENA) | From baseline to 3-month follow-up
  It collects information on emotional and behavioural problems by means of a self-report questionnaire (8 to 12 years old) composed of 134 items where the participant has to choose one option on a five-point scale (Never or almost never to Always or almost always); examples: 'I am told that I interrupt others and that I don't let them talk', 'school is stupid'. The questionnaire evaluates four blocks of scales: I) scales of problems, composed of internalised problems (depression, anxiety, social anxiety and somatic complaints), externalised problems (attention problems, hyperactivity-impulsivity, anger control, aggression and defiant behaviour), II) contextual problems, family problems, problems with the school and with peers, III) scales of vulnerabilities, problems of emotional regulation and IV) scales of personal resources, self-esteem, integration and social competence.
Compassion Scale for Children (CSC) | From baseline to 3-month follow-up
  This questionnaire measures three factors related to compassion: compassion for other people, compassion for oneself and compassion for other living beings. The scale consists of 20 items whose responses employ a 5-point Likert format for responses, where 1 indicates "Never," 2 means "Rarely," 3 represents "Sometimes," 4 indicates "Often," and 5 signifies "Always". The minimum score is 20 points and the maximum is 100, with the higher the score indicating a higher level of compassion.
Academic performance | From baseline to 3-month follow-up
  Each student's academic performance will be assessed by comparing the average grade obtained in all subjects taught in the trimester before and after the intervention.

SECONDARY OUTCOMES:
Qualitative assessment for students | 9 weeks
  Students will answer a short 7-question survey in open-ended format and Likert-type scale that covers aspects such as perceived usefulness, putting into practice what they have learned, benefits and degree of satisfaction with the programme carried out.
Semi-structured global impression interview for teachers | 9 weeks
  At the end of the intervention, a semi-structured interview will be carried out with the tutor of each class, consisting of 9 questions in an open-ended format and Likert-type scale. This interview has been designed by Carlos García Rubio and collaborators (García-Rubio et al. 2019) and collects information on the subjective perception of the feasibility of the intervention, the beneficial and detrimental effects, the general impression and the potential of the intervention.

OTHER OUTCOMES:
Participant age | At baseline
  Age of participants, measured in years.
Course | At baseline
  Course attended by the student.
Gender | At baseline
  Participant's gender

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology and Sociology. Faculty of Education. University of Zaragoza, Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No